CLINICAL TRIAL: NCT02771847
Title: Impact of Comorbidities Among Adolescents Infected Pain Associated With Disorders of the Masticatory System
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 14-PP-14
Record Dates: First submitted 2016-05-10; First posted 2016-05-13 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Masticatory System
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: survey — anonym survey is given to people

SUMMARY:
The pain associated with disorders of the masticatory system (DAM) include pain in the masticatory muscles, temporomandibular joints, or deux.1-5 In terms of frequency, the DAM is the second musculoskeletal disorder most common behind chronic pain in the dos.

Pain associated with DAM not interested adults; they were also observed in adolescents (2-6%) 7 with significant changes in their quality of life.8 The annual incidence of pain associated with DAM is 2.6% among adolescents and 3.9% for adults. 9 half to two-thirds of patients affected by DAM resorted to professional care, and one-third continued to be subjected to moderate pain and incapacity to severe, regardless of treatment given.

Co-morbidities were identified in adults 12-14, children and adolescents with pain related to DAM, the United States and Suède. The most common painful co-morbidities among children and adolescents were headaches, neck, back, limbs or abdomen.

The reasons for the co-existence of DAM with other painful conditions are not well understood. Nevertheless, it has been demonstrated in adults that they contributed to apparition and persistence DAM beyond healing time conventionally predicted; they increased deterioration state health and could complicate significantly the diagnosis and efficacy of treatment.

Co-morbidity is defined as "the simultaneous existence and the occur two or more diseases, medically diagnosed in the same person.

The prevalence of several chronic painful conditions appears to be greater among people of low socioeconomic status compared with those of higher and higher socioeconomic status among women than hommes.

head pain is commonly reported in the general population (46%) The headache prevalence ranges from 9% to 97% among adults and 30% to 94% among Adolescents with DAM.

Women have a higher probability have pain related to DAM (odds ratio (OR) = 2.2, 95% confidence interval (CI): 2.1-2.4) or headache (OR = 2.5, 95% CI: 2.4-2.5) than men. Cross-sectional studies and case-control demonstrated that subjects with DAM-related pain were 1.5 to 8.8 times more likely to have headaches compared to those without pain associated with DAM.

The relationship between headaches and DAM n'est unclear. Both conditions seem to share similar pathophysiological mechanisms that would promote the development of both diseases in a individual. Patients affected by headaches are more likely to develop a DAM? A cohort study showed that adolescents affected by headaches, the chance of developing pain related to DAM was 2.7 times (95% CI: 1.6-4.4) than adolescents without headaches. Conversely, the probability of having headache increases with the number of symptoms according to a relationship of DAM.

Following the results of these studies cited before, it is now necessary to confirm the relationship between headaches and DAM among adolescents.

Neck pain and back are symptoms commonly reported in adults with DAM (35% to 44%). 23 The adults affected by DAM have smaller mobility angles in the cervical and more sensitive points to trapezoids when compared to those without DAM.

Cross-sectional studies and case-control have demonstrated that adult patients with DAM-related pain had 2.6 to 5 times more likely have back pain than individuals without pain related to DAM. Chances pain joint (OR = 4.0, 95% CI: 3.7-4.3) are larger among adults affected by DAM related pain compared to those indemnes. adults affected by DAM-related pain were also more likely to experience neck pain (OR = 4.0 to 7.9).

Adult women affected by DAM-related pain are more likely to have pain in the neck (OR = 1.5; 95% CI: 1.4-1.8) and back (OR = 1.2; 95% CI: 1.2-1.3) compared to hommes a prospective cohort study demonstrated that there was a greater likelihood of pain related to DAM among adolescents affected by back pain compared to those not affected (OR = 3.0, 95% CI: 2.2-6.8) Our study aims to seek more evidence on the supposed relationship between pain related to DAM and sore neck or back in the adolescent population.

The irritable bowel syndrome (CIS; 9% to 16%), interstitial cystitis (17%), and stomach pain (34%) are rated among adults affected by DAM. Adults affected by DAM were 2.7 times (95% CI: 1.4-5.1) more likely to have irritable bowel syndrome than subjects of the same age not affected. teenagers affected by DAM were 1.5 times (95% CI: 1.0- 2.1) over have luck stomach upset that the subjects of the same age unaffected.

ELIGIBILITY:
Inclusion Criteria:

* adolescents between 14 and 16
* agree to complete an anonymous survey

Exclusion Criteria:

-

Ages: 14 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: adolescents in 8 school in Nice
Sampling Method: Non-Probability Sample
Enrollment: 566 (Actual)
Dates: Start 2015-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
number of painful co-morbidities of DAM among adolescents | 12 months
  identification of co-morbidities by survey analyses

SECONDARY OUTCOMES:
number of non-painful co-morbidities of DAM among adolescents | 12 months
  identification of co-morbidities by survey analyses

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No